CLINICAL TRIAL: NCT01345500
Title: Randomized Clinical Trial of a Weight Loss Program in Type 2 Diabetes
Brief Title: UCSD Take Charge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: HealthPartners Institute (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Cheryl Rock, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110463
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Overweight; Obese; Obesity; Diabetic; Type 2 Diabetes
Keywords: Overweight; Obese; Type 2 Diabetic; Diabetes; Weight loss; Physical activity; Diet; Prepackaged meals
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Higher Carbohydrate/Lower Fat Diet (Experimental)
  Interventions: Other: Higher Carbohydrate, Lower Fat Diet
- Lower Carbohydrate/Higher Fat Diet (Experimental)
  Interventions: Other: Lower carbohydrate, Higher fat diet
- Individualized Counseling (Active Comparator)
  Interventions: Other: Individualized Counseling

INTERVENTIONS:
Other: Higher Carbohydrate, Lower Fat Diet — Study participants will receive prepackaged prepared foods as needed to achieve a meal plan, free-of-charge for a 12-month period. The lower fat, higher carbohydrate diet provides 60% energy from carbohydrate, 20% energy from fat, and 20% energy from protein. The diet falls within the range of current dietary recommendations.
  Arms: Higher Carbohydrate/Lower Fat Diet
Other: Lower carbohydrate, Higher fat diet — Study participants will receive prepackaged prepared foods as needed to achieve a meal plan, free-of-charge for a 12-month period. The lower carbohydrate, higher fat diet provides 45% energy from carbohydrate, 35% energy from fat, and 20% energy from protein. The diet falls within the range of current dietary recommendations.
  Arms: Lower Carbohydrate/Higher Fat Diet
Other: Individualized Counseling — Participants assigned to the usual care group will be provided consultation with a research staff dietetics professional, who will provide publicly available print material that describes dietary and physical activity guidelines to promote weight loss and maintenance, at baseline (after randomization) and again at 6 months.
  Arms: Individualized Counseling

SUMMARY:
The purpose of the Take Charge Study is to determine among overweight and obese men and women with type 2 diabetes whether 1) participating in a commercial weight loss program promotes great weight loss and weight loss maintenance at one year compared to usual care conditions and 2) whether there is a differential weight loss response to different dietary macronutrient composition (lower carbohydrate/higher fat diet versus a higher carbohydrate/lower fat).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Type 2 diabetes
* BMI 25-45 kg/m2
* Willing to participate in any of the study diet arms (higher or lower carbohydrate diet or usual care) over a one-year period
* Able to comply with all required study procedures and schedule
* Must live within the San Diego or Minneapolis area

Exclusion Criteria:

* Pregnant, breastfeeding or planning to become pregnant in the next year
* Serious medical condition or psychiatric illness
* History of having an eating disorder, food allergy or food intolerance
* Have food restrictions or requires a special diet
* Objects to frozen, processed or prepackaged foods
* Inability to be moderately physically active
* Currently enrolled in a weight loss program or another diet intervention
* Current use of weight loss medication or supplements
* Planned surgical procedure that can impact the conduct of the study
* Previous surgical procedures for weight reduction
* Does not have own transportation
* Have plans to relocate from area within 1 year
* HbA1C >11%, fasting triglycerides >600 mg/dL, serum creatinine >1.4 mg/dL (women) or 1.5 mg/dL (men) -- to be screened at baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Total weight loss | 1 year
  To test, in a randomized controlled trial, whether participation in a commercial weight loss program promotes greater weight loss and weight loss maintenance at one year in overweight or obese men and women with type 2 diabetes compared to usual care conditions.

SECONDARY OUTCOMES:
Response to macronutrient composition | 1 year
  To examine whether there is a differential weight loss response at 3, 6 and/or 12 months to different dietary macronutrient composition (higher carbohydrate and lower fat versus lower carbohydrate and higher fat) in the weight loss intervention in these overweight or obese men and women with type 2 diabetes.
Biochemical/social outcomes | 1 year
  To describe the effect of participating in the program (vs. usual care) on markers of glycemic control, cardiovascular disease risk, cardiopulmonary fitness, plasma carotenoids, quality of life, and eating attitudes and behaviors. Also to examine whether there is a differential response to different dietary macronutrient composition in the two weight loss intervention groups in selected metabolic factors, lipids and CRP at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - HealthPartners Research Foundation and University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Rock CL, Flatt SW, Pakiz B, Taylor KS, Leone AF, Brelje K, Heath DD, Quintana EL, Sherwood NE. Weight loss, glycemic control, and cardiovascular disease risk factors in response to differential diet composition in a weight loss program in type 2 diabetes: a randomized controlled trial. Diabetes Care. 2014 Jun;37(6):1573-80. doi: 10.2337/dc13-2900. Epub 2014 Apr 23. PMID 24760261